CLINICAL TRIAL: NCT00407303
Title: A Phase I/II Study of Obatoclax Mesylate (GX15-070MS) Administered in Combination With Bortezomib to Patients With Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Brief Title: Safety and Efficacy of Obatoclax Mesylate (GX15-070MS) in Combination With Bortezomib for the Treatment of Relapsed or Refractory Mantle Cell Lymphoma (MCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Gemin X (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GEM012
Record Dates: First submitted 2006-12-01; First posted 2006-12-05 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Mantle-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — obatoclax; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental): 30mg obatoclax, 1.0mg/m2 bortezomib
  Interventions: Drug: Obatoclax mesylate; Drug: Bortezomib
- 2 (Experimental): obatoclax 30 mg, bortezomib 1.3 mg/m2
  Interventions: Drug: Obatoclax mesylate; Drug: Bortezomib
- 3 (Experimental): Obatoclax 45 mg, Bortezomib 1.3 mg/m2
  Interventions: Drug: Obatoclax mesylate; Drug: Bortezomib

INTERVENTIONS:
Drug: Obatoclax mesylate — 30 mg, 45 mg
  Other Names: (GX15-070MS)
Drug: Bortezomib — 1.0mg/m2, 1.3 mg/m2

SUMMARY:
Defects in the apoptotic process can lead to the onset of cancer by allowing cells to grow unchecked when an oncogenic signal is present. Obatoclax is designed to restore apoptosis through inhibition of the Bcl-2 family of proteins, thereby reinstating the natural process of cell death that is often inhibited in cancer cells.

DETAILED DESCRIPTION:
This is a multi-center, open-label, Phase I study of Obatoclax administered in combination with bortezomib in 3-week cycles to patients with relapsed or refractory Mantle Cell Lymphoma. Treatment may be administered on an outpatient basis. No investigational or commercial agents or therapies other than those described herein may be administered with the intent to treat the patients's malignancy. Supportive care measures including those directed at controlling symptoms resulting from Mantle Cell Lymphoma are allowed.

ELIGIBILITY:
Inclusion Criteria:

* Pathological confirmation of Mantle Cell Lymphoma (ML)
* Must have documented relapse or progression following 1 or 2 prior lines of antineoplastic therapy
* Must have normal organ function
* Must have the ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

* No other agents or therapies administered with the intent to treat malignancy
* Patients with prior exposure to obatoclax
* Uncontrolled, intercurrent illness
* Pregnant women and women who are breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2006-10; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Determine the response rate to obatoclax in combination with Bortezomib and characterize the safety profile | 4 weeks to 2 years

SECONDARY OUTCOMES:
Peripheral blood counts; Bone marrow aspirates and biopsies; Transfusion and growth factor requirements | 4 weeks to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean Viallet, MD, Study Director — Gemin X, Inc.
Locations (5):
- United States (5):
  - NW Georgia Oncology Centers, Marietta, Georgia
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Roswell Park Medical Center, Buffalo, New York
  - University of Wisconsin, Madison, Wisconsin